CLINICAL TRIAL: NCT02588989
Title: Fibrosis, Valvular and Ventricular Function in Patients With Transposition of the Great Arteries
Brief Title: Fibrosis, Valvular and Ventricular Function in Patients With TGA
Status: Active, not recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: TGA_function
Record Dates: First submitted 2015-10-22; First posted 2015-10-28 (Estimated); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Transposition of Great Vessels
MeSH Terms: conditions — Transposition of Great Vessels

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Intracellular RNA collection from whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- transposition of the great arteries: Patients with a TGA

SUMMARY:
The aim of this project is to better evaluate the systemic right ventricular (RV) function in patients with transposition of the great arteries (TGA).

DETAILED DESCRIPTION:
Patients with TGA frequently develop supraventricular and ventricular arrhythmia, conduction problems, systemic atrioventricular valve (SAVV) regurgitation, and congestive heart failure (CHF), all at young age. However, there is variation in time of onset of these adverse events. We want to evaluate ventricular and valvular function at rest, markers of RV fibrosis and cardiac reserve.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a TGA
* Informed consent to participate. If the patient is under the age of 18, the assent of the patient and the permission of the parents to participate

Exclusion Criteria:

* Previous double-switch intervention
* Any medical contra-indication for cardiovascular magnetic resonance (CMR) imaging (e.g. pacemaker)
* The presence of exercise-induced arrhythmia, symptomatic myocardial ischemia, a resting systolic blood pressure > 200 mm Hg and/or diastolic blood pressure > 110 mm Hg, New York Heart Association (NYHA) class III or IV, or non-cardiac co-morbidity that could aggravate by exercise
* Additional exclusion criterion for delayed gadolinium enhancement CMR: any medical contra-indication for intravenous gadolinium

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a transposition of the great arteries (TGA)
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | 10 years
  Composite clinical end point

CONTACTS AND LOCATIONS:
Overall Officials: Werner Budts, M.D., Ph.D., Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Jan Bogaert, M.D., Ph.D., Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium